CLINICAL TRIAL: NCT05472389
Title: Neurodevelopmental Impact of Epilepsy on Autonomic Function in Dravet Syndrome
Acronym: AUTONOMIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL22_0370
Record Dates: First submitted 2022-06-16; First posted 2022-07-25 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Dravet Syndrome; Epilepsy
Keywords: Dravet Syndrome; Epilepsy
MeSH Terms: conditions — Epilepsies, Myoclonic; Epilepsy | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients, adults and children, with Dravet Syndrome (Other): An homogenous population of patients with DS. The patients will have a prospective baseline period of 3 to 6 months duration in order to collect seizure frequency. After this period, all patients will then undergo a 24-48 hours video-EEG recordings and a full-night polysomnography
  Interventions: Other: Video-electroencephalography; Other: Blood Samples

INTERVENTIONS:
Other: Video-electroencephalography — All patients will be monitored 24 hours. Whenever possible, duration of the long-term monitoring will be extended to 48 hours, including a second full night polysomnography. These recordings will also allow us to assess sleep architecture and to capture seizures in some patients video , EEEG, EKG, respiration and other polysomnography data will be centralized at Hospices Civils de Lyon. A copy of the EEG-EKG data required to address the objectives related to cardiac features will then be electronically transferred to Partner 2 (Bonn) Evaluation will be performed blind to other data by the Partner 1 (Lyon) for the respiratory data and by the Partner 2 (Bonn) for the EKG data All primary outcomes and secondary outcomes will be assessed with respect to duration of epilepsy and frequency of convulsive seizures during the baseline period.
Other: Blood Samples — Blood samples will be collected at V2 in all patients. A total of seven blood samples of 4 ml each will be collected, including five EDTA and two dry. Samples EDTA plasma and serum will then be prepared after centrifugation. In children < 10 kg, only 5 samples of 4 ml each (22 ml in total), including four EDTA and one dry.

SUMMARY:
Dravet Syndrome (DS) is a severe epileptic encephalopathy, which main cause is mutations of SCN1A, the gene coding for the Nav1.1 voltage-gated sodium channel. DS is characterized by childhood onset, severe cognitive deficit and drug-resistant seizures, including several generalized convulsive seizures per day, frequent status epilepticus and high seizure-related mortality rate. Sudden and unexpected death in epilepsy (SUDEP) represents the major cause of premature deaths. The risk of SUDEP is thus about 9/1000-person-year in comparison with about 5/1000-person-year in the whole population of patients with drug-resistant epilepsies.

Experimental and clinical data suggest that SUDEP primarily result from a postictal central respiratory dysfunction. SUDEP in DS, might be the result of a seizure-induced fatal apnea in a patient who had developed epilepsy-related vulnerability to central autonomic and/or respiratory dysfunction. However, a key clinical issue which remains to be addressed is the temporal dynamics of the onset and evolution of the autonomic vulnerability in these patients. The main clinical risk factor of SUDEP is the frequency of convulsive seizures and the SUDEP risk can vary along the evolution of epilepsy. Although non-fatal seizure-induced ataxic breathing can be observed in patients with DS, whether or not repetition of seizures results in long-term alterations of breathing remains unclear.

In the AUTONOMIC project, it will be investigate in a homogenous population of patients with DS the exact interplay between epilepsy-related cardiac and respiratory alterations on the one hand and the relation between the underlying neurodevelopmental disease, the repetition of seizure per se and these epilepsy-related autonomic alterations on the other hand.

Autonomic functions will be investigated in the inter-ictal period (i.e. in the absence of immediate seizures, Work Package 1 (WP1)) and in the peri-ictal period, i.e. in the immediate time before, during (if possible) and after seizures (WP2). A multicenter cohort will be constituted, allowing to collect the inter-ictal and ictal cardio-respiratory data required in the 2 WP. The study will be sponsored by the Lyon's University Hospital.

Patients will be recruited over a period of 24 months in one of the three participating clinical center. All patients will first enter in a prospective baseline period of 3 to 6 months duration in order to collect seizure frequency. After this period, all patients will then undergo a 24-48 hours video-EEG recordings as part of the routine clinical care. The monitoring will also include a full-night polysomnography. This patients will be eligible for inclusion in an extension follow-up study will monitor vital status every year in order to investigate long-term mortality, including SUDEP.

The AUTONOMIC project will provide important results which will pave the way to develop and eventually validate therapeutic intervention to prevent SUDEP. By deciphering the exact interplay between epilepsy-related cardiac and respiratory alterations on the one hand and the relation between the underlying neurodevelopmental disease, the repetition of seizure per se and these epilepsy-related autonomic alterations on the other hand, the project will primarily deliver clinically relevant biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Children (> 2 years and < 18 years) and adult patients (< 60 years) with established diagnosis of Dravet Syndrome
* Adults protected by a guardianship or curatorship
* Diagnosis of Dravet syndrome will be confirmed by PI of each study center based on medical history, type of seizures, EEG data and results of genetic testing
* No restriction related to the seizure frequency
* Patient (or patient's parents or legal representative) who gave its written informed consent to participate to the study
* At least one of the parents and/or legal representative understanding and speaking national language
* Written consent form signed by both parents
* Absence of known current pregnancy and breastfeeding
* Patient affiliated to its national health care system

Exclusion Criteria:

* Patients (children or adults) unable to tolerate at least 24 hours of video-EEG recordings (behavioural problems resulting in technical issues for appropriate EEG recordings)
* Patients with congenital heart or lung disease
* Patients with congenital abnormalities or diseases, other than the epilepsy, which could interfere with sleep
* Subject in exclusion period of another study

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2035-09-11 (Estimated)

PRIMARY OUTCOMES:
Respiratory primary outcome for the inter-ictal period : measure of the total duration of central sleep apnea (sec/min/hours) during total sleep time over a 24-hour period | Data collected during 24 hours of video-EEG.
  Total duration of central sleep apneas during total sleep time over a 24-hour period at Visit 2
Cardiac primary outcome for the inter-ictal period: ratio's calculation of root mean square of successive differences (RMSSD) during wakefulness and sleep | Data collected during 24 hours of video-EEG at Visit 2
  Ratio of root mean square of successive differences (RMSSD) during wakefulness and sleep
Respiratory primary outcome for the peri-ictal period :occurrence's measure of post-convulsive central apnea during the 30 sec to 10 min after the end of convulsive seizure | Between 30 seconds and 10 minutes after the end of the convulsive seizure at Visit 2
  Occurrence of post-convulsive central apnea
Cardiac primary outcome for the peri-ictal period : measurement of ictal QTc-lengthening ≥60 ms during the 30 sec to 10 min after the end of convulsive seizure | Between 30 seconds and 10 minutes after the end of the convulsive seizure at visit 2
  Ictal QTc-lengthening, ≥60 ms

SECONDARY OUTCOMES:
Respiratory secondary outcomes for the inter-ictal period : calculation of central apnea index | Data collected during 24 hours of video-EEG.
  Central apnea index: Total number of central apneas divided by total sleep time over a 24-hour period.
Respiratory secondary outcomes for the inter-ictal period : measurement of Total duration of central sleep apneas during each sleep stage over a 24-hour period (sec/min) | Data collected during 24 hours of video-EEG.
  Total duration of central sleep apneas during each sleep stage over a 24-hour period.
Respiratory secondary outcomes for the inter-ictal period : calculation of Obstructive Apnea Hypopnea Index | Data collected during 24 hours of video-EEG.
  Obstructive Apnea Hypopnea Index: Total number of obstructive apneas, obstructive hypopneas, and mixed apneas divided by total sleep time) over a 24-hours period.
Respiratory secondary outcomes for the inter-ictal period : measurement of total duration of periods with tcCO2 >50 mmHg during total sleep time over a 24-hour period (sec/min) | Data collected during 24 hours of video-EEG.
  Total duration of periods with tcCO2 >50 mmHg during total sleep time over a 24-hour period
Respiratory secondary outcomes for the inter-ictal period : measurement of total duration of periods with pulse oximetry <90% during total sleep time over a 24-hour period | Data collected during 24 hours of video-EEG.
  Total duration of periods with pulse oximetry <90% during total sleep time over a 24-hour period
Cardiac secondary outcomes for the inter-ictal period calculation of standard deviation of R-R intervals | Data collected during 24 hours of video-EEG.
  Standard deviation of R-R intervals over the time period (SDNN) during sleep and during wakefulness.
Cardiac secondary outcomes for the inter-ictal period : percentage's calculation of consecutive R-R intervals differing by > 50 milliseconds (pNN50) during sleep and during wakefulness (%) | Data collected during 24 hours of video-EEG.
  Percentage of consecutive R-R intervals differing by > 50 milliseconds (pNN50) during sleep and during wakefulness.
Cardiac secondary outcomes for the inter-ictal period : calculation of ratio between the low frequency and high frequency spectrum (LF/HF ratio) of the RR-interval. (Hz) | Data collected during 24 hours of video-EEG.
  Ratio between the low frequency (LF, 0.04-0.15 Hz) and high frequency (HF, 0.15-0.4 Hz) spectrum (LF/HF ratio) of the RR-interval
Cardiac secondary outcomes for the inter-ictal period : analysis of ration of sleep to wakefulness for each HRV variables | Data collected during 24 hours of video-EEG.
  Ratio of sleep to wakefulness for each HRV variable. HRV features are determined during a period of at least 10 min in artifact-free recording during wakefulness at rest and sleep stage N3 and REM sleep.
Cardiac secondary outcomes for the inter-ictal period : measurement of the evolution of Heart Rate Variability variable during hyperventilation procedure | Data collected during 24 hours of video-EEG.
  Evolution of HRV variable during hyperventilation procedure.
Cardiac secondary outcomes for the inter-ictal period : analysis of T wave alternans (V) | Data collected during 24 hours of video-EEG.
  T wave alternans (TWA). TWA is the beat-to-beat variation of morphology and amplitude of the ST segment or T wave and mirrors temporo-spatial heterogeneity of cardiac repolarization
Respiratory secondary outcomes for the peri-ictal period : duration's measurement of post-convulsive central apnea (sec/min) | Between 30 seconds and 10 minutes after the end of the convulsive seizure.
  Duration of PCCA in patients in whom it occurs
Respiratory secondary outcomes for the peri-ictal period : occurrence's measurement of ataxic breathing | Between 30 seconds and 10 minutes after the end of the convulsive seizure.
  Occurrence of ataxic breathing (i.e. irregular breathing rhythm) in the post-ictal period
Respiratory secondary outcomes for the peri-ictal period : occurrence and duration's measurement of period of tcCO2 >50 mm Hg in the post-ictal period (sec/min) | Between 30 seconds and 10 minutes after the end of the convulsive seizure.
  Occurrence and duration of period of tcCO2 >50 mm Hg in the post-ictal period
Respiratory secondary outcomes for the peri-ictal period : measurement of Delay between the end of the seizure and recovery of oxygen saturation (SpO2) ≥90% (sec/min) | Between 30 seconds and 10 minutes after the end of the convulsive seizure.
  Delay between the end of the seizure and recovery of oxygen saturation (SpO2) ≥90%
Respiratory secondary outcomes for the peri-ictal period : measurement of desaturation nadir | Between 30 seconds and 10 minutes after the end of the convulsive seizure.
  Desaturation nadir in the immediate aftermath of a convulsive seizure
Cardiac secondary outcomes for the peri-ictal period : occurrence's measurement of peri-ictal asystole | Between 30 seconds and 10 minutes after the end of the convulsive seizure.
  Occurrence of peri-ictal asystole (sinus arrest of ≥3s)
Cardiac secondary outcomes for the peri-ictal period : occurrence's measurement of peri-ictal bradycardia | Between 30 seconds and 10 minutes after the end of the convulsive seizure.
  Occurrence of peri-ictal bradycardia (<2nd HR percentile for age; average of three consecutive RR intervals)
Cardiac secondary outcomes for the peri-ictal period : measurement of all Heart Rate Variability (HRV) | Between 30 seconds and 10 minutes after the end of the convulsive seizure.
  All HRV measures described in the inter-ictal period will also be collected and analyzed in the 15 minutes immediately following the end of the seizure (because of movement artefacts HRV measures are not reliable during the course of convulsive seizures)
Cardiac secondary outcomes for the peri-ictal period : measurement of T wave alternans | Between 30 seconds and 10 minutes after the end of the convulsive seizure.
  T wave alternans (TWA) in the 15 minutes immediately following the end of the seizure
Additional features : measurement of the the postictal generalized EEG suppression (V) | All measurements will take place during hospitalization for 24/48 hours at Visit 2 after the baseline period
  Total duration of the postictal generalized EEG suppression, defined as lack of detectable EEG activity >10 in amplitude on all leads
Additional features : measurement of the total duration of the postictal coma (sec/min/hours) | During hospitalization for 24/48 hours at Visit 2 after the baseline period
  Total duration of the postictal coma, defined as the delay between the end of the seizure and the recovery of consciousness assessed by the ability to meet one single verbal command (handshake).
Additional features : measurement of the total duration of the postictal immobility (sec/min/hours) | During hospitalization for 24/48 hours at Visit 2 after the baseline period
  Total duration of the postictal immobility, defined as the delay between the end of the seizure and the first spontaneous movement of the patient, as assessed on the video recording.

CONTACTS AND LOCATIONS:
Locations (4):
- Department of Paediatrics and Paediatric Neurology, Antwerp University Hospital, Edegem, Belgium
- France (2):
  - HFME Hospices Civils de Lyon, Bron, Rhone
  - Hôpital Neurologique Pierre Wertheimer Hospices Civils de Lyon, Bron, Rhone
- Klinik und Poliklinik für Epileptologie, Universitätsklinikum, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No